CLINICAL TRIAL: NCT03085342
Title: Evaluation of Hepatic Fibrosis on Multiparametric MRI Including Portal Flow Measurement Using Dual-input Software: Preliminary Study
Brief Title: Evaluation of Hepatic Fibrosis on Multiparametric MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2015-2993
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cirrhosis; Hepatitis
Keywords: liver; fibrosis; MRI
MeSH Terms: conditions — Fibrosis; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver MRI (Experimental): Liver MRI including noncontrast (precontrast) flow measurement, DCE, DWI using multiple b-values, MRE and MR fat quantification.
  Interventions: Diagnostic Test: Liver MRI

INTERVENTIONS:
Diagnostic Test: Liver MRI — Multiparametric Liver MRI including following sequences: DCE, DWI, MRE, precontrast flow measurement, fat quantification.

SUMMARY:
As cirrhosis progresses, alteration of hemodynamics develops and decreased portal flow is often observed. Since direct measurement of portal pressure (HVPG) is invasive, non-invasive methods have drawn a lot of attention. MRI is one of the non-invasive methods and it is able to provide multiparametric data in one examination. Herein, we evaluate hepatic fibrosis with different stage using multiparametric MRI with emphasis on portal flow measurement.

ELIGIBILITY:
Inclusion Criteria:

* chronic liver disease (viral hepatitis, alcoholic hepatitis, or other...)
* Or transplant recipient for viral hepatitis and on anti-viral agent medication
* AND scheduled for liver resection, biopsy or transient elastography
* AND signed informed consent

Exclusion Criteria:

* younger than 18 years
* any contra-indication for contrast-enhanced MRI
* pregnant or nursing women
* biliary obstruction
* unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
hepatic fibrosis stage | 1 month after MRI
  F0-1 vs. F2-4 using multiparametric MRI

SECONDARY OUTCOMES:
presence of varix | 1 month after MRI
  presence of esophageal or gastric varices using multiparametric MRI
comparison of portal flow measurement | 1 month after MRI
  comparison of portal flow measurement using DCE and precontrast flow measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No